CLINICAL TRIAL: NCT01726218
Title: Enhancing Stroke Recovery Through Cortical Stimulation: The Role of the Ipsilateral Motor Cortex in Executing Movements With Increasing Demand on Precision
Brief Title: Role of Ipsilateral Motor Cortex in Executing Movements With Increasing Demand on Precision
Acronym: RIMC
Status: Completed | Type: Observational
Sponsor: Cathrin Buetefisch (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Cathrin Buetefisch, Dr Cathrin Buetefisch, M.D., PhD, Emory University
Organization: Emory University (Other)
Other Study IDs: IRB00048694; R56NS070879-01 (NIH); RIMCR56 (Other: Other)
Record Dates: First submitted 2012-03-29; First posted 2012-11-14 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Stroke
Keywords: Stroke; Physical Medicine & Rehabilitation; Neurology; Neurophysiology; Neuroscience; Transcranial Magnetic Stimulation (TMS)
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stroke patients
- Healthy Control

SUMMARY:
It is well known that the motor area of one hemisphere of the brain (motor cortex) controls the movement of the opposite of the body. However, it is not clear whether as the movement becomes more complicated, the motor cortex of both hemispheres of the brain are involved. Currently the role of the motor cortex on the same side of the body (referred to as ipsilateral motor cortex) in hand performance remains controversial. The investigators demonstrated previously in healthy subjects that transiently lowering the activity of ipsilateral motor cortex improved the performance of the opposite hand. What is not know are the mechanisms involved in these changes of behavior. Transcranial magnetic stimulation (TMS) is a device that allows the non- invasive stimulation of the brain. When brain is stimulated repetitively at a very low rate and low intensity for about 15 minutes, the stimulated brain area becomes less active. This effect lasts 10 minutes and is called a "transient artificial lesion" as it mimicks the effects of transiently interfering with the function of the stimulated brain area. In the present study the investigators will conduct experiments using repetitive TMS to downregulate the activity of the motor area as in previous experiments and measures its effect on activity of motor cortex of both hemispheres. The investigators will study healthy subjects. It would be important to understand the effects in more detail for the design of treatment strategies in patients after stroke, which will be a topic of future studies.

ELIGIBILITY:
Inclusion Criteria for Stroke Patients:

* Age 18-80
* Single cerebral ischemic infarction one month prior to entering study
* Affecting only one hemisphere as defined by MRI of the brain
* At the time of cerebral infarct a motor deficit of hand of Medical Research Council Scale for Muscle Strength (MRC) of < 4- of wrist and finger extension/flexion movement
* Fugl Meyer score > 27/66 (motor domain, upper extremity)
* Ability to operate joystick at largest target level
* No other neurological disorder
* No intake of Central Nervous System (CNS) active drugs
* Ability to give informed consent
* Ability to meet criteria of inclusion experiment
* No major cognitive impairment

Inclusion Criteria for Healthy Subjects:

* Age 55-80 years with no neurological or psychiatric diseases
* Normal neurological examination
* Normal MRI of the brain
* Normal neuropsychological testing
* No intake of CNS active drugs that interfere with data collection
* No contraindication to TMS
* Ability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 Stroke patients with 15 in each group based on location of stroke 50 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2015-03-26 (Actual); Study Completion 2015-03-26 (Actual)

PRIMARY OUTCOMES:
Define key parameters that contribute to contralesional M1 reorganization following stroke | Up to six months post-stroke

CONTACTS AND LOCATIONS:
Overall Officials: Cathrin Buetefisch, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Wischnewski M, Edwards L, Revill KP, Drake D, Hobbs G, Buetefisch CM. Intensity-Dependent Effects of Low-Frequency Subthreshold rTMS on Primary Motor Cortex Excitability and Interhemispheric Inhibition in Elderly Participants: A Randomized Trial. Neurorehabil Neural Repair. 2025 Jan;39(1):58-73. doi: 10.1177/15459683241292615. Epub 2024 Oct 27. PMID 39462433